CLINICAL TRIAL: NCT04102436
Title: A Phase II Study Using the Administration of Autologous T-Cells Engineered Using the Sleeping Beauty Transposon/Transposase System to Express T-Cell Receptors Reactive Against Mutated Neoantigens in Patients With Metastatic Cancer
Brief Title: Non-Viral TCR Gene Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty with availability of GLP-grade reagents for manufacturing.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190143; 19-C-0143
Record Dates: First submitted 2019-09-24; First posted 2019-09-25 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Endocrine/Neuroendocrine; Non-Small Cell Lung Cancer; Breast Cancer; Gastrointestinal/Genitourinary Cancers; Ovarian Cancer
Keywords: Adoptive Cell Therapy; Cell Therapy; Immunotherapy; Gene Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Urogenital Neoplasms; Ovarian Neoplasms | interventions — fludarabine; Cyclophosphamide; aldesleukin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Sleeping Beauty (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + Sleeping Beauty Transposed PBL + high- or low-dose aldesleukin.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Aldesleukin; Biological: Sleeping Beauty Transposed PBL

INTERVENTIONS:
Drug: Fludarabine — Days -7 to -3: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days.
Drug: Cyclophosphamide — Days -7 and -6: Cyclophosphamide 60 mg/kg/day x 2 days IV in 250 mL D5W infused simultaneously with mesna 15 mg/kg/day over 1 hour x 2 days.
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg or 72,000 IU/kg (based on total body weight) IV over 15 minutes approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 10 doses).
Biological: Sleeping Beauty Transposed PBL — Day 0: Cells are to be infused at a dose not to exceed 1.5e11 in 400 mL intravenously on the Patient Care Unit over 20-30 minutes or as clinically determined by an investigator for patient safety (between 2-4 days after the last dose of fludarabine).

SUMMARY:
Background:

A person s white blood cells can be modified in a lab to recognize certain changes in their tumor. Many of these cells are collected from the person, modified, then given back to the person. This may help treat some cancers.

Objective:

To learn if a person s white blood cells modified with T-cell receptors can cause solid tumors to shrink.

Eligibility:

People ages 18-70 who have cancer of the gastrointestinal tract, genitourinary tract, ovary, breast, or lung that has spread, or who have glioblastoma.

Design:

Participants will be screened and have their cells prepared for treatment in another protocol.

Participants will be hospitalized one week before treatment. They will stay approximately 3 - 4 weeks after treatment.

Participants will get the modified white blood cells and chemotherapy through an IV catheter, which is a small plastic tube inserted in a vein.

Participants will take drugs by mouth to prevent infection. They will receive filgrastim as a shot or injection under the skin.

Participants will have tests before, during, and after treatment:

Heart, blood, and urine tests

Chest X-ray

Physical exam

Scans: They will lie in a machine that takes pictures of the body.

Possible apheresis: The participant s blood is removed through a needle in an arm. The blood goes through a machine that removes the white blood cells. The rest of the blood is returned through a needle in the other arm.

Participants will have visits about 6 and 12 weeks after treatment. If they are responding to treatment, they will then have visits every 3-6 months for 3 years. Then they will join another study and be followed about 12 more years.

DETAILED DESCRIPTION:
Background:

* The administration of autologous tumor infiltrating lymphocytes (TIL) can mediate complete, durable regressions in 20-25% of patients with metastatic melanoma. Recent studies have shown that these TIL predominantly recognize unique mutated neoantigens expressed by the cancer not shared by other melanomas.
* Administration of bulk autologous TIL to patients with a variety of other solid cancers, including cancers of the gastrointestinal tract and genitourinary tract, have little if any therapeutic impact.
* Recent studies in the Surgery Branch, NCI, have shown that TIL from non-melanoma solid cancers can also contain T-cells reactive against non-shared unique mutated neoantigens expressed in the cancer. The frequency of these T-cells is very low (often < 0.1%) and it is thus difficult to isolate and grow mutation reactive T-cells to levels required for effective therapy.
* In several patients with chemo-refractory metastatic epithelial cancers, we were able to grow an enriched population of neoantigen reactive TIL and administration of these cells mediated several partial regressions of metastatic disease and one complete regression of all metastatic breast cancer now lasting more than 3 years.
* We have now developed approaches to identify these rare neoantigen reactive T-cells from common non-melanoma cancers, to isolate their T-cell receptors (TCR), and to genetically engineer autologous peripheral blood lymphocytes (PBL) using the Sleeping Beauty system to express these TCRs with high efficiency. The neoantigen TCR gene- modified cells can recognize and destroy the autologous cancer in vitro.
* We are now proposing a clinical protocol to treat patients with refractory solid cancers using the adoptive transfer of autologous PBL transposed with genes encoding TCRs that recognize unique mutated neoantigens expressed by the cancer.

Objective:

-To determine the rate of objective response (using RECIST v1.1 criteria) of patients with solid cancers who receive autologous PBL that have been genetically modified with genes encoding TCRs that recognize mutated neoantigens in the autologous cancer using the Sleeping Beauty system.

Eligibility:

Patients who are age greater than or equal to 18 years and less than or equal to 70 years must have:

* Measurable solid cancer with at least one lesion that is resectable for TIL generation with minimal morbidity plus at least one other lesion that can be measured that falls into one of four cohorts: (1) gastrointestinal and genitourinary, (2) breast and ovarian, (3) non- small cell lung cancer (NSCLC), and (4) glioblastoma. Metastatic disease is required for Cohorts 1-3 but not for Cohort 4.
* Evaluable solid cancer that has recurred following standard chemotherapy or standard erapy OR therapy has been declined
* Adequate organ function
* No allergies or hypersensitivity to cyclophosphamide, fludarabine, or aldesleukin.
* No concurrent major medical illnesses or any form of immunodeficiency

Design:

* Patients will undergo resection or biopsy to obtain tumor for generation of autologous TIL cultures. Patients will be entered into four cohorts that include (1) gastrointestinal and genitourinary tract cancers, (2) breast and ovarian cancers, (3) non-small cell lung cancer (NSCLC), and (4) glioblastomas. Exome sequencing and often RNA Seq will be performed to identify the mutations expressed in the patient s cancer. Multiple autologous TIL cultures will be grown and tested for reactivity against mutations from the autologous tumor using assays we have developed that involve the exposure of autologous antigen presenting cells to long peptides containing the mutation or tandem mini genes encoding the mutation.
* T-cell cultures with reactivity against mutations will be identified and the individual TCRs that recognize the mutation will be synthesized and used to transfect the TCR into patient s autologous PBL using the Sleeping Beauty system.
* Transposed autologous PBL will then be expanded to large numbers using our standard rapid expansion protocol and administered to the patient following a non-myeloablative lymphodepleting regimen.
* All patients will receive a non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine. Patients will then receive the infusion of autologous transposed PBL and begin high-dose aldesleukin (720,000 IU/kg IV every 8 hours for up to 10 doses).
* Clinical and immunologic response will be evaluated approximately 4-6 weeks after cell infusion and periodically thereafter.
* It is anticipated that approximately one patient per month will enroll into the trial for each of the four histologic groups. Thus, accrual of up to 4 x 50=200 total evaluable patients may be completed in approximately 2-4 years. In order to allow for a small number of inevaluable patients the accrual ceiling will be set to 210.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with histologically confirmed solid cancer that falls into one of four cohorts:

  * Gastrointestinal and genitourinary (Cohort 1),
  * Breast and ovarian (Cohort 2),
  * Non-small cell lung cancer (NSCLC), NSCLC includes but is not limited to squamous cell carcinoma, adenosquamous carcinoma or adenocarcinomas (Cohort 3),
  * Glioblastoma (Cohort 4)
* Patients must have evaluable or measurable disease per RECIST 1.1 with at least one lesion that is resectable for TIL generation with minimal morbidity plus at least one other lesion that can be measured. Metastatic disease is required for Cohorts 1-3 but is not required for Cohort 4.
* Patients must have:

  * previously received standard systemic therapy for their advanced cancer and have been either non-responders or have recurred, specifically:

    * Patients with metastatic colorectal cancer must have received oxaliplatin or irinotecan (or similar agents)
    * Patients with breast and ovarian cancer must be refractory to first-line treatments
    * Patients with lung cancer must have received at least one platinum-based chemotherapy regimen and at least one FDA-approved targeted treatment (when appropriate)
    * Patients with glioblastoma must have progression of disease after radiotherapy (including patients that undergo surgery for recurrent disease and are rendered NED). This includes recurrent GBM after receiving all standard first-line treatment, including surgery (if feasible due to neurosurgical and neuro- anatomical considerations) and adjuvant radiotherapy +/- chemotherapy. OR
  * declined standard treatment
* For Cohorts 1-3: Patients with 3 or fewer brain metastases that are < 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for one month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
* For Cohort 3: Patients must have documented FEV1 > 60% predicted.
* Age greater than or equal to 18 years and less than or equal to 70 years.
* For Cohorts 1-3: Clinical performance status of ECOG 0 or 1.
* For Cohort 4: Patients must have Karnofsky performance status of greater than or equal to 60.
* The effects of study treatment on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) at time of study entry, for the duration of treatment and up to 4 months after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Serology

  * Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus may be less responsive to the experimental treatment and more susceptible to its toxicities.)
  * Seronegative for active hepatitis B, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
* Hematology

  * ANC > 1,000/mm^3 without the support of filgrastim
  * WBC greater than or equal to 3,000/mm^3
  * Platelet count greater than or equal to 100,000/mm^3
  * Hemoglobin > 8.0 g/dL. Subjects may be transfused to reach this cut-off.
* Chemistry

  * Serum ALTlAST less than or equal to 5.0 x ULN
  * Serum creatinine less than or equal to 1.6 mgldL
  * Total bilirubin less than or equal to 1.5 mg/dL, except in patients with Gilbert s Syndrome, who must have a total bilirubin < 3.0 mg/dL.
* More than four weeks must have elapsed since completion of any prior systemic therapy and enrollment.

Note: Patients may have undergone minor surgical procedures or limited field radiotherapy (with the exception of patients with glioblastoma) within the four weeks before enrollment, as long as any related major organ toxicities have recovered to less than or equal to grade 1.

* For Cohort 3: More than two weeks must have elapsed since any prior palliation for major bronchial occlusion or bleeding and enrollment, and patient s toxicities must have recovered to less than or equal to grade 1.
* For Cohort 4: Patients must be at least four weeks from radiation therapy. Additionally, patients must be at least six weeks from nitrosoureas, four weeks from temozolomide, three weeks from procarbazine, two weeks from vincristine and four weeks from last bevacizumab administration. Patients must be at least four weeks from other cytotoxic therapies not listed above and two weeks for non-cytotoxic agents (e.g., interferon) including investigative agents. Patient s toxicities must have recovered to less than or equal to grade 1.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Willing to sign a durable power of attorney.
* Subjects must be co-enrolled on protocol 03-C-0277.

EXCLUSION CRITERIA:

* Pregnant women are excluded from this study because study treatment s potential for teratogenic or abortifacient effects is unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with study therapy, breastfeeding should be discontinued if the mother is treated on this trial.
* Concurrent systemic steroid therapy, except for patients with glioblastoma (Cohort 4).
* Active systemic infections requiring anti-infective treatment, coagulation disorders or any other active or uncompensated major medical illnesses.
* For Cohort 3: Any major bronchial occlusion or bleeding not amenable to palliation.
* For Cohort 4: Clinically significant hemorrhagic or ischemic stroke, including transient ischemic attacks and other central nervous system bleeding in the preceding six months that were not related to glioma surgery.

Note: History of prior intratumoral bleeding is not an exclusion criterion; however, patients with a history of prior intratumoral bleeding will need to undergo a non- contrast head CT to exclude acute bleeding.

* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune- competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
* History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, or aldesleukin.
* History of coronary revascularization or ischemic symptoms.
* Documented LVEF less than or equal to 45% tested in patients:

  * Age greater than or equal to 65 years
  * With clinically significant atrial and/or ventricular arrhythmias, including but not limited to: atrial fibrillation, ventricular tachycardia, second- or third-degree heart block, or have a history of ischemic heart disease and/or chest pain.
* Documented FEVl less than or equal to 50% predicted tested in patients with:

  * A prolonged history of cigarette smoking (greater than or equal to 20 pack-year smoking history within the past two years).
  * Symptoms of respiratory dysfunction.
* Clinically significant patient history which in the judgment of the Principal Investigator (PI) would compromise the patients ability to tolerate high-dose aldesleukin.
* Patients who are receiving any other investigational agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 and 12 weeks after cell infusion, then every 3 months x3, then every 6 months x 2 years, then per PI discretion
  Percentage of patients who have a clinical response to treatment (objective tumor regression)

SECONDARY OUTCOMES:
Phenotypic and functional characteristics of PBL | 2-4 years post cell infusion
  Patient PBL will be obtained from whole blood and then evaluated for function and phenotype.
Safety and tolerance | 6 weeks (+/- 2 weeks) following administration of the cell product
  Using standard CTCAE 5.0
Immune monitoring | 6 weeks (+/-2 weeks) following administration of the cell product
  Will consist of quantifying T-cells reactive with HLA-matched tumor cells using established techniques such as intracellular FACS, cytokine release assays, and ELISpot assays.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Deniger DC, Switzer K, Mi T, Maiti S, Hurton L, Singh H, Huls H, Olivares S, Lee DA, Champlin RE, Cooper LJ. Bispecific T-cells expressing polyclonal repertoire of endogenous gammadelta T-cell receptors and introduced CD19-specific chimeric antigen receptor. Mol Ther. 2013 Mar;21(3):638-47. doi: 10.1038/mt.2012.267. Epub 2013 Jan 8. PMID 23295945
- [Background] Ivics Z, Hackett PB, Plasterk RH, Izsvak Z. Molecular reconstruction of Sleeping Beauty, a Tc1-like transposon from fish, and its transposition in human cells. Cell. 1997 Nov 14;91(4):501-10. doi: 10.1016/s0092-8674(00)80436-5. PMID 9390559
- [Background] Maiti SN, Huls H, Singh H, Dawson M, Figliola M, Olivares S, Rao P, Zhao YJ, Multani A, Yang G, Zhang L, Crossland D, Ang S, Torikai H, Rabinovich B, Lee DA, Kebriaei P, Hackett P, Champlin RE, Cooper LJ. Sleeping beauty system to redirect T-cell specificity for human applications. J Immunother. 2013 Feb;36(2):112-23. doi: 10.1097/CJI.0b013e3182811ce9. PMID 23377665
- [Derived] Levy PL, Gros A. Fast track to personalized TCR T cell therapies. Cancer Cell. 2022 May 9;40(5):447-449. doi: 10.1016/j.ccell.2022.04.013. Epub 2022 May 9. PMID 35537408
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0143.html